CLINICAL TRIAL: NCT00662675
Title: A Randomized Double-blind (Withdrawal) Phase 3 Study to Evaluate the Efficacy and Tolerability of Pancrelipase MT Capsules Compared With Placebo in the Treatment of Subjects With Cystic Fibrosis-dependent Exocrine Pancreatic Insufficiency
Brief Title: A Study of the Efficacy and Tolerability of Pancrelipase Microtablet (MT) Capsules for the Treatment of Cystic Fibrosis-dependent Exocrine Pancreatic Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014719
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2010-03-17 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Exocrine Pancreatic Insufficiency; Steatorrhea; Malabsorption Syndromes; Cystic Fibrosis
Keywords: Exocrine pancreatic insufficiency; Steatorrhea; Malabsorption syndromes; Cystic fibrosis; Pediatrics; Adult; Pancrelipase
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Steatorrhea; Malabsorption Syndromes; Cystic Fibrosis | interventions — MT 21

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 001 (Experimental): Pancrease MT 10.5 or MT 21 Pancrease MT capsules for maximum dose of 10 000 lipase units / Kg / day
  Interventions: Drug: Pancrease MT 10.5, or MT 21
- 002 (Experimental): Placebo for Pancrease MT 10.5 or MT 21 Capsules with Pancrease MT excipients without the active enzymes
  Interventions: Drug: Placebo for Pancrease MT 10.5 or MT 21

INTERVENTIONS:
Drug: Pancrease MT 10.5, or MT 21 — Pancrease MT capsules for maximum dose of 10,000 lipase units / Kg / day
  Arms: 001
Drug: Placebo for Pancrease MT 10.5 or MT 21 — Capsules with Pancrease MT excipients without the active enzymes
  Arms: 002

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of oral pancrelipase MT in the treatment of adult and pediatric/adolescent cystic fibrosis (CF) patients with clinical symptoms of exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind withdrawal, multicenter study to evaluate the effectiveness of pancrelipase MT capsules compared with placebo in the treatment of adult (>18 to 60 years of age) and children/adolescent (7 to <18 years of age) patients with CF and who require pancreatic enzyme replacement therapy (PERT) to control clinical symptoms of EPI and steatorrhea (excess fat in the feces). The study has 3 phases: a screening phase, an open-label (run-in) phase, and a double-blind withdrawl phase. The study including the screening phase will be approximately 28 days in length. In the screening phase, patients will begin a high-fat diet and will take pancrelipase MT10.5 or MT21 capsules (or a combination of both) orally with meals (or snacks) to optimize digestion based on clinical signs and symptoms. In the open-label phase patients will continue taking their optimal dose of study drug. After a minimum of 3 days in the open-label treatment phase, an inpatient 72-hour stool collection period for fecal fat determination will be performed. Patients with a coefficient of fat absorption (COA)-fat of 80% or greater who have completed at least 6 days on a controlled high-fat diet will be eligible for the double-blind withdrawal phase of the study and will be randomly assigned to receive placebo or pancrelipase MT. After a minimum of 1 day on double-blind treatment and with the presence of deteriorating clinical signs and symptoms, patients will be admitted to the clinic to begin a second 72-hour inpatient stool collection period. Effectiveness evaluations will be performed throughout the study and consist of stool collection for determination of COA-fat and coefficient of protein absorption (COA-protein), stool diary, nutrition worksheet, and Clinical Global Impression-Severity of illness (CGI-S), Clinical Global Impression-Change (CGI-C), and Global Assessment of Change (GAC) scales. Signs and symptoms exhibited during the study will be monitored and will include the presence or absence of diarrhea, abdominal pain, nausea, vomiting, bloating, and a description of stool changes. Safety will be montitored during the study by evaluating adverse events and findings from clinical laboratory tests, vital signs measurements, and physical examinations. The study hypothesis is that the study drug will be more effective than placebo as measured by the change in the coefficient of fat absorption (COA-fat) in adults and pediatric/adolescent patients with EPI secondary to CF. Pancrelipase MT10.5 or MT21 capsules (or a combination of both) will be taken orally with meals (or snacks) within the recommended ranges of pancreatic enzyme therapy as recommended by the CF Foundation and up to a maximum 10,000 lipase units per kilogram [kg] per day. All patients will take pancrelipase MT for 6 days in the screening phase and for approximately 6 to 10 days in the open-label phase; patients will take pancrelipase MT or placebo for 4 to 7 days in the double-blind phase.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of CF documented by sweat chloride results (>60 mmol/L) and require pancreatic enzyme replacement therapy (PERT) to control clinical symptoms of EPI (nausea, vomiting, bloating, diarrhea, and abdominal pain) with a history of excess fat in the feces
* Have documentation of an abnormal COA-fat and a fecal elastase result of <100 micrograms fecal elastase/gram stool
* Must be on a stable diet and dose of pancreatic enzyme supplementation that has provided satisfactory symptom control for at least the past 1 month

Exclusion Criteria:

* No extreme physical wasting with loss of weight and muscle mass
* No severe, acute, or chronic pulmonary disease unrelated to complications of CF
* No worsening of pulmonary disease in past 30 days
* No use of drugs known to affect blood uric acid concentrations (e.g., aspirin, diflunisal, allopurinol, probenecid, thiazide diuretics, phenylbutazone, sulfinpyrazone)
* No known congenital (present at birth) abnormalities of the gastrointestinal tract, heart, or liver
* No distal intestinal obstruction syndrome (DIOS)

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (11):
- United States (10):
  - Long Beach, California
  - Los Angeles, California
  - Orlando, Florida
  - Louisville, Kentucky
  - Las Vegas, Nevada
  - Long Branch, New Jersey
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
- Vancouver, British Columbia, Canada

REFERENCES:
- See also: A randomized double-blind (withdrawal) Phase 3 study to evaluate the efficacy and tolerability of PANCREASE MT capsules compared with placebo in the treatment of subjects with cystic fibrosis-dependent exocrine pancreatic insufficiency — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=77&filename=CR014719_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial (screening) dose of PANCREASE MT was based on the average dose of pancreatic enzyme replacement therapy (PERT) taken for the 3 days immediately before entry into the study in combination with a high-fat diet. This PERT was continued until all screening test results were received and the subject met all inclusion/exclusion criteria.
Groups:
- Placebo: Matching placebo capsules taken by mouth per meal or snack
- PANCREASE MT: Pancrease MT 10.5 or MT 21 capsules taken by mouth per meal or snack
Period: Overall Study
Arm/Group | Placebo | PANCREASE MT
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PANCREASE MT | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (11.58) | 24 (13.44) | 23.7 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in the Coefficient of Fat Absorption (COA-fat Percent)
Description: Change in the coefficient of fat absorption (percent COA-fat) from the 72-hour inpatient period in the open-label phase to the 72-hour period inpatient period in the double-blind (withdrawal) phase.
Time Frame: 72-hours stool collection in the open-label phase to the end of 72-hours stool collection in the double-blind withdrawal phase.
Population: Intent-to-Treat (ITT)
Measure: Mean (Standard Deviation); unit: percentage COA-fat
Arm/Group | Placebo | PANCREASE MT
Number analyzed (Participants) | 20 | 20
percentage COA-fat | -34.1 (23.03) | -1.5 (5.88)
Statistical Analysis 1: Comparison: Placebo vs PANCREASE MT; The power calculation was based on the assumption that the true mean difference between the active and the placebo group was 31.2% with a common standard deviation of 22.6% using a 2-sided, 2-sample, t-test with a 5% significance level; Test type: Superiority or Other; p < 0.001, ANCOVA; The p-value is from ANCOVA model with treatment as a factor and baseline percent COA-fat as a covariate

2. Secondary Outcome: Change in Percent COA-Protein (Nitrogen)
Description: The change in percent COA-protein from the stool collection period in double-blind phase to open-label phase
Time Frame: as for outcome 1
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage COA-protein
Arm/Group | Placebo | PANCREASE MT
Number analyzed (Participants) | 20 | 20
percentage COA-protein | -26.5 (15.3) | 1.3 (4.71)
Statistical Analysis 1: Comparison: Placebo vs PANCREASE MT; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value is from ANCOVA model with treatment as a factor and baseline percent COA-protein(nitrogen) as a covariate

3. Secondary Outcome: Percent of Patients Reporting Clinical Signs and Symptoms of Exocrine Pancreatic Insufficiency (EPI) During the Double-Blind Phase
Description: Percent of patients reporting nausea, vomiting, bloating, diarrhea, oily/greasy stools, and abdominal pain signs and symptoms reported as Adverse events during the double-blind phase.
Time Frame: Entire 7 days double-blind phase
Population: ITT
Measure: Number; unit: Percent of participants
Arm/Group | Placebo | PANCREASE MT
Number analyzed (Participants) | 20 | 20
Percent of participants
  % of subjects with at least one EPI symptoms | 55 | 20
  % of subjects with Abdominal pain | 30 | 15
  % of subjects with Bloating | 15 | 5
  % of subjects with Diarrhea | 20 | 0
  % of subjects with Greasy stools | 15 | 0
  % of subjects with Vomiting | 0 | 5

ADVERSE EVENTS:
Time Frame: During the 7 days double-blind withdrawal phase
Arm/Group | Placebo | PANCREASE MT
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | PANCREASE MT (N=20)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1
Abnormal faeces (Gastrointestinal disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less